CLINICAL TRIAL: NCT01703234
Title: FGF-23 and Endothelial Dysfunction in Diabetic Proteinuric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Mahmut Ilker Yilmaz, Assoc.Prof., Gulhane School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: GATARAMFGF232012
Record Dates: First submitted 2012-10-04; First posted 2012-10-10 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Proteinuria; Diabetic Nephropathy; Chronic Kidney Disease
Keywords: FGF-23 , ramipril, endothelial dysfunction
MeSH Terms: conditions — Proteinuria; Diabetic Nephropathies; Renal Insufficiency, Chronic | interventions — Ramipril

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Ramipril (Experimental)
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Ramipril — ramipril 10 mg/day during 3 months

SUMMARY:
There is no data about the effects of Renin angiotensin system blockage (RAS) on FGF23 and ADMA levels in diabetic patients with proteinuria. The aim of this study was to find out whether the beneficial effects of RAS blockage in diabetic proteinuria has any relation with the alteration of ADMA and FGF-23 levels. We searched for the effects of ACE inhibitor ramipril on the clinical and laboratory parameters of diabetic patients with proteinuria.

DETAILED DESCRIPTION:
In recent years, diabetic nephropathy, which may lead to dialysis treatment, is the most prevalent underlying disease of people in developed countries. A wide range of studies have been carried out, from various points of view, to understand the progress of renal dysfunction in diabetic nephropathy. The endogenous nitric oxide synthase (NOS) inhibitor asymmetric dimethylarginine (ADMA) is elevated in patients with chronic kidney disease (CKD) and may have a role in the cardiovascular mortality and morbidity of these patients. In diabetic nephropathy, high ADMA levels were related to progression of diabetic nephropathy.

Fibroblast growth factor 23 (FGF-23) is a primary regulator of renal phosphate excretion. FGF23 is inversely associated with the GFR, a relationship underlying a fundamental mechanism for maintaining serum phosphate constancy during CKD progression. Such an adaptation may have deleterious trade-offs because, independently of serum phosphate, high FGF23 signals a high risk of death in ESRD patients. Some studies showed that there is a relationship between FGF-23 levels and proteinuria in CKD patients.

There is no data about the effects of Renin angiotensin system blockage (RAS) on FGF23 and ADMA levels in diabetic patients with proteinuria. The aim of this study was to find out whether the beneficial effects of RAS blockage in diabetic proteinuria has any relation with the alteration of ADMA and FGF-23 levels. We searched for the effects of ACE inhibitor ramipril on the clinical and laboratory parameters of diabetic patients with proteinuria.

The study 'Effect of Renin Angiotensin System Blockade on the Fas Antigen (CD95) and Asymmetric Dimethylarginine (ADMA) Levels in Type-2 Diabetic Patients With Proteinuria' has been previously registered to ClinicalTrials.gov (Identifier:NCT00893425). The serum samples of the above study will be used in order to measure the FGF23 levels in this study. Therefore the eligibility criteria and the study design is similar to the previous study (Identifier:NCT00893425).

The patients who were non-obese (BMI<30kg/m2), non dyslipidemic (total cholesterol <200mg/dl, Triglyceride<150mg/dl), and free of cardiovascular events (negative medical history, negative ECG findings) were investigated for enrollment. CKD stage 1 patients older than 18 years of age and willing to participate to the study were screened. From the 231 patients with established type 2 diabetes mellitus, 126 had proteinuria and/or hypertension (24 h protein excretion 1-2 g/day, systolic blood pressures ≥140mmHg and/or diastolic blood pressures ≥ 90 mmHg, respectively). All cases were first referrals and at the time of the study all were off treatment. Patients with history of coronary artery disease, smokers and those taking statins or renin-angiotensin blockers were excluded because of the effect of these factors on endothelial dysfunction. Of 126 screened patients 78 met the study criteria and were included in this study. The duration of proteinuria and diabetic nephropathy after initial diagnosis was not known.

The exclusion criteria were as follows: A)Nephrotic syndrome, B)coronary heart disease (patients with ischemic ST-T alterations and voltage criteria for LVH on electrocardiogram, and with history of revascularization or myocardial infarction), C) elevated liver enzymes (AST or ALT levels ≥ 40U/L) and D) renal failure (serum creatinine levels > 1.3 mg/dl). In order to evaluate the effect of RAS blockade on FGF 23 concentrations, patients with proteinuria were given an ACE inhibitor (ramipril 10 mg/day) for 12 weeks. The effect of RAS blockade on insulin sensitivity and proteinuria was also investigated.

After the intervention period, blood samples were obtained for assay of FGF-23 concentrations, HbA1c , and insulin resistance scores (HOMA-IR).

Urine samples were also collected over a 24-hour period to determine the degree of proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 1 patients
* Older than 18 years of age
* Type 2 Diabetic patients
* Proteinuria

Exclusion Criteria:

* History of coronary artery disease
* Smokers
* Taking statins or renin-angiotensin blockers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Flow Mediated Dilatation

SECONDARY OUTCOMES:
FGF-23

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane School of Medicine, Ankara, Turkey (Türkiye)